CLINICAL TRIAL: NCT07375589
Title: Exploratory Study on the Efficacy and Safety of LED Low-Intensity Red Light for Controlling Myopia Progression in Children and Adolescents
Brief Title: LED Low-Intensity Red Light for Myopia Control in Youth: Efficacy and Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Beijing Airdoc Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLED-2025
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-04

CONDITIONS: Myopia; Ametropia
Keywords: Myopia
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LED Red light: 1.6 mW/twice daily (Experimental)
  Interventions: Device: Red light treatment with 1.6mW LED light source
- LED Red light: 0.001 mW/twice daily (Sham Comparator)
  Interventions: Device: Red light treatment with 0.001mW LED light source

INTERVENTIONS:
Device: Red light treatment with 1.6mW LED light source — In addition to using a powered single vision glasses lens (SVS) to correct distance refraction, the subjects underwent two red light treatments using a 1.6mW LED light source therapy device from Monday to Friday, each treatment was 3 minutes, and the interval was 4 hours.
  Arms: LED Red light: 1.6 mW/twice daily
Device: Red light treatment with 0.001mW LED light source — In addition to using a powered single vision glasses lens (SVS) to correct distance refraction, subjects were treated with red light twice from Monday to Friday using a 0.001mW LED light source therapy instrument, each time for 3 minutes, with an interval of 4 hours.
  Arms: LED Red light: 0.001 mW/twice daily

SUMMARY:
The purpose of this clinical trial was to investigate the efficacy and safety of repetitive low-intensity single-wavelength red light from an LED light source in controlling myopia progression in children and adolescents.

DETAILED DESCRIPTION:
Myopia is the most prevalent ocular condition among children and adolescents worldwide. In recent years, optical interventions for myopia prevention and control have gained increasing attention, with low-intensity red light (wavelength: 650 nm) emerging as a promising therapeutic approach. Clinical studies have preliminarily demonstrated the efficacy of repeated low-level red light (RLRL) therapy in slowing myopia progression in pediatric populations. Existing research has primarily utilized semiconductor laser diodes due to their high monochromaticity and concentrated beam intensity. However, concerns persist regarding the safety of red light irradiation in clinical myopia management. The primary risks include potential damage to intraocular structures from prolonged or high-intensity exposure, coupled with the high cost of laser-based systems, which limits their widespread adoption.

In contrast to laser sources, light-emitting diodes (LEDs) operate via non-thermal mechanisms and deliver significantly lower energy output, mitigating the risk of thermal or photochemical tissue damage. Investigating the efficacy and safety of low-intensity red LED light for controlling myopia progression in children and adolescents is therefore of critical scientific and clinical importance.This study aims to evaluate the effectiveness and safety of repeated low-intensity, single-wavelength (650 nm) red LED light therapy in slowing axial elongation in children aged 8-12 years over a 3-month treatment period. Participants will receive RLRL therapy at home under parental supervision in addition to wearing single-vision spectacles, following a standardized protocol. Key outcome measures, including axial length (AL), visual acuity, cycloplegic spherical equivalent refraction (SER), intraocular pressure (IOP), slit-lamp biomicroscopy, optical coherence tomography (OCT), and optical biometry, will be assessed at baseline and at 1-week, 1-month, and 3-month follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 8-12 years old
2. Simple myopia: equivalent spherical lens ≤ -0.5D and > -6.0D after any cycloplegia, astigmatism ≤ 2.5D, anisometropia ≤ 1.5D
3. The best corrected visual acuity in one eye is 0.8 and above
4. Normal fundus, or only leopard-shaped fundus
5. Sign informed consent and be able to participate in the study

Exclusion Criteria:

1. Rule out hereditary myopia
2. The subject has other congenital eye diseases, such as congenital cataract, congenital glaucoma, etc
3. Presence of strabismus or other binocular vision abnormalities
4. refractive media opacity: corneal opacity, cataract or intraocular lens surgery
5. There are eye diseases that affect retinal function
6. Children who had used or were using orthokeratology, atropine and other myopia control measures could be enrolled after stopping treatment for three months
7. There are other systemic disease abnormalities
8. Other reasons that the research doctor considers unsuitable for inclusion in the project

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Subjects in the intervention group received red light treatment with 1.6mW LED light source during 3 months | 1 week，1 ,3months
  Subjects in the intervention group received red light treatment with 1.6mW LED light source for 3 months, and the change of axial length was compared with the increase of axial length in the blank group

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China